CLINICAL TRIAL: NCT02066571
Title: A Phase II, Double-Blind, Placebo-Controlled, Crossover Study to Assess Clinical Benefit and Safety of Droxidopa in the Treatment of Parkinson's Disease
Brief Title: Study to Assess the Clinical Benefit and Safety of Droxidopa in Parkinson's Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Peter LeWitt MD, M.D., Henry Ford Health System
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: LeWitt01; IND 119340 (Other: FDA)
Record Dates: First submitted 2014-02-18; First posted 2014-02-19 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Parkinson's Disease; Freezing of Gait; Cognitive Ability, General
Keywords: Parkinson's disease; Freezing of gait; Gait
MeSH Terms: conditions — Parkinson Disease | interventions — Droxidopa; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- droxidopa, then sugar pill (Other): Droxidopa will be titrated over a 2-week period up to 300 mg twice daily (600 mg total daily dose). Subjects will be titrated to highest tolerated dose and will continue on that dose for two weeks. Then, the subject will start sugar pills.
  Interventions: Drug: Droxidopa; Drug: sugar pill
- sugar pill, then droxidopa (Other): Subject will be be on sugar pill for 5 weeks (4 weeks of placebo treatment and one week of wash-out or sugar pills). Then, droxidopa will be titrated over 2 week period up to 300 mg twice daily (600 mg total daily dose). Subjects will be titrated to highest tolerated dose and will continue on that dose for two weeks.
  Interventions: Drug: Droxidopa; Drug: sugar pill

INTERVENTIONS:
Drug: Droxidopa — Droxidopa will be supplied in 100 and 200 mg pill sizes. The proposed dosing is 100mg twice daily at baseline, then titrate to 200 mg twice daily at day 7 and then titrate to 300mg twice daily at day 14. Subjects will stay on the 600mg daily for 2 weeks. Total exposure 28 days of study drug.
Drug: sugar pill — Sugar pill or placebo will be supplied in pill sizes matched to droxidopa formulation. The study titration will be the same. Sugar pills will be used for 5 weeks during the study.
  Other Names: placebo

SUMMARY:
Since droxidopa has been approved in Japan for treating freezing of gait in Parkinson's disease patients, this is to confirm and further investigate the safety and efficacy using a similar dose. The possible beneficial effects on cognition in mildly cognitively impaired Parkinson's disease patients will also be tested, since this problem in Parkinson's disease may be associated with decreased brain synthesis of norepinephrine (a neurotransmitter associated with multiple brain functions).

During this 11 week study, droxidopa will be slowly titrated up to 600 mg daily. Walking and freezing of gait will be evaluated and rated. Cognitive functions will be evaluated by a computer-based program.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent to participate in the study
* Diagnosed with probable levodopa-responsive idiopathic PD (meeting United Kingdom PD Brain Bank diagnostic criteria), and receiving levodopa therapy for this disorder. Other PD medications can also be used.
* Must have AT LEAST ONE of below two criteria:

  1. At least 3 months incidence of typical freezing of gait symptoms, occurring while levodopa is otherwise providing an "on" mobility state (including at least one of the following Freezing of Gait patterns: start hesitancy, freezing at making turns or when passing through a doorway, spontaneous freezing during continued walking, or Freezing of Gait related to a simultaneous mental or physical activity) OR
  2. Have a screening score between 22 and 26 (inclusive) on the Montreal Cognitive Assessment

Exclusion Criteria:

* Taking direct acting vasoconstriction agent (i.e. ephedrine or midodrine). Subjects taking vasoconstrictor agents such as ephedrine or midodrine must stop taking these drugs at least 2 days or 5 half-lives (whichever is longer) prior to their baseline visit
* Taking anti-hypertensive medication for the treatment of hypertension. Anti-hypertensive medication taken at night to prevent supine hypertension will be allowed
* Changing dose or frequency of PD medication within 2 weeks of baseline
* Use of cognitive-enhancing medications (donepezil, galantamine, rivastigmine, tacrine, or memantine), catechol-O-methyltransferase inhibitors (tolcapone or entacapone), anticholinergic drugs, or antipsychotic drugs (including quetiapine or clozapine).
* Known or suspected alcohol or substance abuse within 1 year (e.g. DSM-IV definition of alcoholism)
* Past or current history of chronic severe hypertension (with repeated findings of BP 150/90 mmHg in the supine or standing position)
* Symptomatic coronary artery disease, severe congestive heart failure (NYHA Class 3 or 4)
* Unable to remain off any effective Freezing of Gait medications for 12 hrs prior to Evaluation visits)
* Women who are pregnant, lactating, or plan to become pregnant during the course of this study
* Women of child bearing potential who are not using two methods of contraception (at least one barrier, i.e. condom) with their partner.
* Male subjects who are sexually active with a woman of child bearing potential and not using two methods of contraception (at least one barrier, for example, condom)
* A history of closed angle glaucoma;
* Active (in the last 6 months) atrial fibrillation or, in the investigator's opinion, any other significant cardiac arrhythmia that should preclude the subject from this trial
* History of myocardial infarction or unstable angina
* Congestive heart failure (NYHA Class 3 or 4)
* Diabetes insipidus, insulin-dependent diabetes mellitus, or diabetic neuropathy
* In the investigator's opinion, any other significant systemic illness
* Known or suspected malignancy (other than basal cell carcinoma)
* Known gastrointestinal illness or other gastrointestinal disorder that may, in the investigator's opinion, affect the absorption of study drug
* Any major surgical procedure within 30 days of the baseline visit
* Currently receiving any investigational drug or have received an investigational drug within 30 days of the baseline visit
* In the investigator's opinion, clinically significant abnormalities on clinical examination or laboratory testing that should preclude the subject from this trial.
* Findings from suicidality screening that are compatible with risk for suicide

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-04 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in freezing of gait symptoms using Freezing of Gait Questionnaire | 4 weeks
  Evaluate the effect of droxidopa on freezing of gait symptoms using the Freezing of Gait Questionnaire completed by patients. All measures will be performed at baseline and after two and four weeks of study medication.
Change from baseline in cognitive testing | 4 weeks
  Battery of cognitive testing is performed. All measures will be performed at baseline and after two and four weeks of study medication.

SECONDARY OUTCOMES:
Change in measurement of freezing of gait | 4 weeks
  Videotaped evaluations quantifying the number of episodes of freezing of gait and their severity will be rated using the Observed Freezing of Gait scale. The Timed Up and Go test will evaluate the effect of droxidopa on PD symptoms. The effect of droxidopa treatment on gait features of stride, swing time variability, and gait asymmetry will be analyzed. All measures will be performed at baseline and after two and four weeks of study medication.
Change in the incidence of falls | 4 weeks
  Videotaped evaluations quantifying the number of fall episodes will be rated using the Observed Freezing of Gait scale. The Timed Up and Go test will evaluate the effect of droxidopa on PD symptoms and freezing of gait. The effect of droxidopa on falls will be analyzed using the GaitRite system.
  All measures will be performed at baseline and after two and four weeks of study medication.
Change in signs and symptoms of Parkinson's disease | 4 weeks
  The UPDRS (Unified Parkinson's Disease Rating Scale) will be performed at baseline and after 2 and 4 weeks on study drug for each arm.
Number of participants with serious and non-serious adverse events | up to 11 weeks
  Safety of droxidopa will be evaluated based on the occurrence of treatment emergent adverse events with specific evaluation of blood pressure, heart rate , ECG, suicidality, and laboratory findings across the study

CONTACTS AND LOCATIONS:
Overall Officials: Peter LeWitt, M.D., Principal Investigator — Henry Ford Health System
Locations (2):
- United States (2):
  - Rush University Medical Center, Chicago, Illinois
  - Henry Ford Hospital, West Bloomfield, West Bloomfield, Michigan